CLINICAL TRIAL: NCT04038229
Title: Biopsychosocial Model for a Multidisciplinary Perioperative Care Pathway in Patients Undergoing Posterior Spinal Fusion Surgery for Adolescent Idiopathic Scoliosis
Brief Title: Multidisciplinary Perioperative Care Pathway in Adolescents Undergoing Posterior Spinal Fusion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Davina Wildemeersch, Principle investigator, University Hospital, Antwerp
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EC19/14/183
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Analgesia; Scoliosis Idiopathic; Surgery; Postoperative Pain
Keywords: enhanced recovery pathway; analgesia; tele-monitoring; biopsychosocial evaluation
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Prospective derived data from children and adolescents undergoing spinal fusion due to idiopathic scoliosis
- Enhanced recovery pathway (Experimental): Children and adolescents undergoing spinal fusion due to idiopathic scoliosis using the pre -per and postoperative enhanced recovery protocol
  Interventions: Other: Enhanced recovery pathway

INTERVENTIONS:
Other: Enhanced recovery pathway — The applied protocol include psychological screening for yellow flags, preoperative gabapentin, peroperative multimodal preemptive management and postoperative holistic evaluation short -and long term
  Arms: Enhanced recovery pathway

SUMMARY:
Posterior Spinal fusion (PSF) is one of the most invasive orthopedic surgical procedures in children and adolescents, often characterized by extensive tissue trauma, and severe postoperative pain. In addition to pain, the postoperative period is complicated by the side effects of opioids such as nausea and vomiting, itching and sedation. Various studies have shown that pain in the direct postoperative phase is an important determinant for development of chronic post-surgical pain.

The consequences of untreated acute pain are known and can also contribute to chronification in pain.

DETAILED DESCRIPTION:
Surgical correction of adolescent idiopathic scoliosis (AIS) is indicated for severe deformity. Posterior Spinal fusion (PSF) for AIS is one of the most invasive orthopedic surgical procedures in children and adolescents, often characterized by a large surgical incision, extensive tissue trauma, risk of blood loss, longer operating times and severe postoperative pain. In addition to pain, the postoperative period is complicated by the side effects of opioids such as nausea and vomiting, itching and sedation. All of this can, along with under-treatment of postoperative pain, be an important delaying factor in postoperative recovery and rehabilitation with a late hospital discharge and increased patient dissatisfaction. Various studies have shown that pain in the direct postoperative phase is an important determinant for development of chronic post-surgical pain.

The consequences of untreated pain are known and can also contribute to chronification in pain.

The incidence of chronic post-surgical pain after scoliosis fusion is 22% at 6 months and 11-15% at 1 to 5 years postoperatively. It is therefore important to minimize the pain during the first postoperative days. Untreated pain in patients is far from benign with significant negative short and long term consequences with accompanying reduction in rehabilitation duration, sleep quality of life. To date, there is no scientific evidence that some analgesic policy is superior, making adequate and safe pain relief and associated anti-emetic therapy after PSF a challenge makes for all healthcare providers involved.

ELIGIBILITY:
Inclusion Criteria:

* approved written informed consent by parent or legal representative
* idiopathic adolescent scoliosis
* planned for elective surgery: posterior spinal fusion

Exclusion Criteria:

* other types of scoliosis
* chronic opioid usage (more than 3 months)
* known unstable psychiatric medical condition

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain | From admission postoperative anesthesia care unit (PACU) up to 3 months postoperatively
  Evaluation of pain at rest and during mobilization using 11 point numeric rating scale daily during hospital admission and is continued after discharge up to 3 months postoperatively

SECONDARY OUTCOMES:
evaluation of opioid-related side effect | From admission postoperative anesthesia care unit (PACU) up to 3 months after surgery
  Evaluation of opioid-related side effect as nausea, vomiting and pruritus
sleep | From admission postoperative anesthesia care unit (PACU) up to 3 months after surgery
  Subjective sleep score using 11 point numeric rating scale
daily activity | From admission postoperative anesthesia care unit (PACU) up to 3 months after surgery
  Subjective activity score using 11 point numeric rating scale
mobility | From day of surgery until hospital discharge (approximately 7 days)
  Daily mobility assessment by attending physiotherapist on 4 point scale

OTHER OUTCOMES:
State-Trait anxiety Inventory (STAI) | 3 times: one to two weeks before planned surgery, 4 weeks after surgery and at 12 weeks after surgery
  evaluation of state and trait characteristics by the STAI questionnaire, via a patient specific online platform
Multidimensional Pain Inventory (MPI, Part 1) | 3 times: one to two weeks before planned surgery, 4 weeks after surgery and at 12 weeks after surgery
  Screening for pain and psychosocial aspects
Child and Adolescent Social and Adaptive Scale (CASAFS) | 3 times: one to two weeks before planned surgery, 4 weeks after surgery and at 12 weeks after surgery
  Screening for pain and psychosocial aspects
Childhood Depression Inventory (CDI-2) | 3 times: one to two weeks before planned surgery, 4 weeks after surgery and at 12 weeks after surgery
  screening for depression
Pain Response Inventory (PRI) | 3 times: one to two weeks before planned surgery, 4 weeks after surgery and at 12 weeks after surgery
  screening for pain coping

CONTACTS AND LOCATIONS:
Overall Officials: Guy Hans, MD, PhD, Study Chair — University Hospital, Antwerp
Locations (1):
- University hospital Antwerp, Edegem, Antwerp, Belgium